CLINICAL TRIAL: NCT01310465
Title: The Effect of Zoledronic Acid to Bone Fusion and Bone Metabolism of Patients With Lumbar Degenerative Disease After Lumbar Interbody Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Jian Dong, Department of Orthopedics of Zhongshan Hospital of Fudan University,
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FudanU-0457034
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-01

CONDITIONS: Image Changes of Lumbar Fusion; Bone Turnover Markers; Bone Mineral Density
MeSH Terms: interventions — Zoledronic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Three days postoperatively, patients in this group are given one infusion of zoledronic acid intravenously.
  Interventions: Drug: zoledronic acid
- Placebo Comparator (Placebo Comparator): Three days postoperatively, patients in this group are given one infusion of sodium chloride intravenously.
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: zoledronic acid — zoledronic acid, 5mg(100ml), intravenous, one time at three days postoperatively
  Arms: Experimental group
Drug: sodium chloride — sodium chloride, 100ml, intravenous, one time at three days postoperatively
  Arms: Placebo Comparator

SUMMARY:
Many patients who have lumbar degenerative disease suffer from osteoporosis or reduced bone mass or low bone mineral density. Among patients with lumbar degenerative disease, some need fusion surgery. But conditions of osteoporosis or low bone mineral density slow down the rate of bone fusion, reduce the success of bone fusion, and ultimately affect the overall effectiveness of surgery. Zoledronic acid is an effective anti-osteoporotic. Many researchers dispute if zoledronic acid can promote the healing of long bone fractures. But few researchers focus on the effect of zoledronic acid to lumbar fusion. In this study, we select patients with lumbar degenerative disease who have had lumbar interbody fusion surgery. Three days postoperatively, the patients were randomized to either one infusion of zoledronic acid or sodium chloride intravenously. We follow all these patients for 6 months. During this time, we detect bone metabolism and bone fusion of these patients. At last, we can tell if zoledronic acid can modify bone metabolism and promote bone fusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar degenerative disease who have had lumbar interbody fusion surgery
* Age 50-70 years old
* Willing to sign informed consent

Exclusion Criteria:

* Application of strontium ranelate, sodium fluoride or parathyroid hormone
* Application of bisphosphonates more than 8 weeks during 2 years preoperatively
* Suffering from bone fracture during 3 months preoperatively
* Urinary creatinine clearance rate less than 35mL/min
* Serum calcium concentrations greater than 2.75mmol/L or less than 2.00mmol/L
* Pregnancy or breast-feeding women
* Suffering from cancer or other diseases that may be expected to live less than a year

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital of Fudan university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Colon-Emeric C, Nordsletten L, Olson S, Major N, Boonen S, Haentjens P, Mesenbrink P, Magaziner J, Adachi J, Lyles KW, Hyldstrup L, Bucci-Rechtweg C, Recknor C; HORIZON Recurrent Fracture Trial. Association between timing of zoledronic acid infusion and hip fracture healing. Osteoporos Int. 2011 Aug;22(8):2329-36. doi: 10.1007/s00198-010-1473-1. Epub 2010 Dec 9. PMID 21153021